CLINICAL TRIAL: NCT04963582
Title: Does LI4 Acupuncture Provide an Effective Analgesia During Intrauterine Device
Brief Title: LI4 Acupuncture for Analgesia in Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Pınar Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08.06.2021/30
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: IUD Insertion Complication; Acute Pain
Keywords: IUD insertion; Acupuncture; Pain management; Acute pain
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Case-controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Experimental): Bilateral LI4 acupuncture is administered before IUD insertion. Pain perception is evaluated by 10 points rated VAS after completion of the procedure.
  Interventions: Procedure: Acupuncture
- Control Group (No Intervention): IUD insertion is proceeded without any intervention. Pain perception is evaluated by 10 points rated VAS after completion of the procedure.

INTERVENTIONS:
Procedure: Acupuncture — LI4 is located on the dorsum of the hand, midway between the 1st and 2nd metacarpal bones, approximately in the middle of the 2nd metacarpal bone on the radial side. Acupuncture is practiced by using 0,25x25mm sized needles. LI4 point is punctured perpendicularly 2cm in the direction of the palm center.
  Arms: Acupuncture Group

SUMMARY:
Pain during IUD insertion is substantially psychologic in origin, responds extremely well to non-pharmacologic interventions. Considering the fact that acupuncture is a modality exerting both psychologic and physiologic effects, the authors presume that acupuncture administration before IUD insertion may have positive effects on pain control. From this point of view, the aim of this study to investigate the effects of LI4 acupuncture administered shortly before IUD insertion on pain perception and discomfort of the women.

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are one the most preferred, most effective and reversible contraceptive methods with long term effects. The major drawback of women for IUD use is the pain anticipation during insertion of the device.

Studies using visual analog scale (VAS) demonstrated that pain perception during IUD insertion varied between 2-7 score. Surprisingly there are only limited number of studies on pain management during IUD insertion which is an ambulatory and out-patient gynecologic procedure. Besides the results of present studies contradict with each other. As a result, a standardized protocol is lacking for pain management in IUD insertion [1]. Currently, most of the IUDs are administered in Community Health Centers (CHC) in our country and no modality for pain control is applied before or after IUD insertion. In case of necessity intramuscular or oral analgesic drugs are prescribed.

In a long-standing review on the basics of this issue, it is concluded that the cervical component of pain perception during IUD insertion is psychologic rather than pathologic, is un-responsive to oral non-steroidal anti-inflammatory drugs and could be deducted via psyche-prophylactic methods. similar results were presented with studies undertaken In the advancing years. A recent study demonstrated that verbal inspiration techniques were as effective as oral tramadol for pain management in IUD insertion. Additionally, the effects of anticipation of pain on perception of pain is essential as well. Because in a large scale study, the results showed that one point increments in the VAS for anticipated pain resulted in an increase of pain perception by 19,7%. Therefore, the fact that psychologic, biologic, cognitive, behavioral, emotional and social factors interfere with pain perception is well-known and it is recommended by clinicians that these factors should be taken into consideration in processes of selecting modalities for pain management.

Scientists research for the mechanism of pain control that acupuncture provides. Acupuncture is extremely effective in autonomic nerve regulation. Also, crucial effects of afferent information within somatic nerve fibers on autonomic functions were demonstrated on experimental and clinical studies. Acupuncture relies on biology based physiologic and psychologic mechanisms. It causes both the secretion of oxytocin and endogen opioids that induce functional changes in various organ systems and rhythmic changes in vulnerable tissues via the stimulation of receptors or nerve fibers.

Acupoint LI4 is the most intensely studied, hte most preferred for analgesia and is the most used acupoint in routine daily practice. Studies on pain management in cases of chest tube pain, dental pain or multiple sclerosis were undertaken using LI4.

ELIGIBILITY:
Inclusion Criteria:

* Women who wish to use IUD as contraception and who refer to Community Health Center for the procedure of IUD insertion.

Exclusion Criteria:

* Women who use anti-coagulant drugs or who have blood diseases.
* Women with dermatologic lesions on the area of LI4 point location.
* Women with previously diagnosed neurologic diseases.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Pain perception | At the 3rd minute after IUD insertion is completed
  Pain perception is measured by using 10-point rated Visuel Analog Scale. Zero point in the scale refers to no pain whereas 10 points refers to worst pain experienced by the patient.
Pain perception | At the 10th minute after IUD insertion is completed
  Pain perception is measured by using 10-point rated Visuel Analog Scale. Zero point in the scale refers to no pain whereas 10 points refers to worst pain experienced by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Erdoğan, MD, Principal Investigator — Niğde Ömer Halisdemir University Midwifery Department
Locations (1):
- Community Health Center, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miles SM, Shvartsman K, Dunlow S. Intrauterine lidocaine and naproxen for analgesia during intrauterine device insertion: randomized controlled trial. Contracept Reprod Med. 2019 Sep 10;4:13. doi: 10.1186/s40834-019-0094-0. eCollection 2019. PMID 31516731
- [Result] Bracken J, Graham CA. Young women's attitudes towards, and experiences of, long-acting reversible contraceptives. Eur J Contracept Reprod Health Care. 2014 Aug;19(4):276-84. doi: 10.3109/13625187.2014.917623. Epub 2014 Jun 2. PMID 24882426
- [Result] Dijkhuizen K, Dekkers OM, Holleboom CA, de Groot CJ, Hellebrekers BW, van Roosmalen GJ, Janssen CA, Helmerhorst FM. Vaginal misoprostol prior to insertion of an intrauterine device: an RCT. Hum Reprod. 2011 Feb;26(2):323-9. doi: 10.1093/humrep/deq348. Epub 2010 Dec 15. PMID 21159683
- [Result] Ngo LL, Ward KK, Mody SK. Ketorolac for Pain Control With Intrauterine Device Placement: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):29-36. doi: 10.1097/AOG.0000000000000912. PMID 26241253
- [Result] Daykan Y, Battino S, Arbib N, Tamir Yaniv R, Schonman R, Klein Z, Pomeranz J, Pomeranz M. Verbal analgesia is as good as oral tramadol prior to intrauterine device (IUD) insertion, among nulliparous women: A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2021 Mar;258:443-446. doi: 10.1016/j.ejogrb.2020.09.019. Epub 2020 Sep 16. PMID 33187752
- [Result] Abu-Zaid A, Alshahrani MS, Albezrah NA, Miski NT, Abuzaid M, Aboudi SA, Baredwan A, Almadhi N, Baradwan A, Alomar O, Salem H, A Al-Badawi I, Baradwan S. Vaginal dinoprostone versus placebo for pain relief during intrauterine device insertion: a systematic review and meta-analysis of randomised controlled trials. Eur J Contracept Reprod Health Care. 2021 Oct;26(5):357-366. doi: 10.1080/13625187.2021.1891411. Epub 2021 Mar 11. PMID 33691549
- [Result] Lopez LM, Bernholc A, Zeng Y, Allen RH, Bartz D, O'Brien PA, Hubacher D. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2015 Jul 29;2015(7):CD007373. doi: 10.1002/14651858.CD007373.pub3. PMID 26222246
- [Result] Goldstuck ND. Pain reduction during and after insertion of an intrauterine contraceptive device. Adv Contracept. 1987 Mar;3(1):25-36. doi: 10.1007/BF01849250. PMID 3630817
- [Result] Origoni M, Leone Roberti Maggiore U, Salvatore S, Candiani M. Neurobiological mechanisms of pelvic pain. Biomed Res Int. 2014;2014:903848. doi: 10.1155/2014/903848. Epub 2014 Jul 8. PMID 25110704
- [Result] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Result] Hunter TA, Sonalkar S, Schreiber CA, Perriera LK, Sammel MD, Akers AY. Anticipated Pain During Intrauterine Device Insertion. J Pediatr Adolesc Gynecol. 2020 Feb;33(1):27-32. doi: 10.1016/j.jpag.2019.09.007. Epub 2019 Sep 26. PMID 31563628
- [Result] Dina B, Peipert LJ, Zhao Q, Peipert JF. Anticipated pain as a predictor of discomfort with intrauterine device placement. Am J Obstet Gynecol. 2018 Feb;218(2):236.e1-236.e9. doi: 10.1016/j.ajog.2017.10.017. Epub 2017 Nov 8. PMID 29079143
- [Result] Andersson S, Lundeberg T. Acupuncture--from empiricism to science: functional background to acupuncture effects in pain and disease. Med Hypotheses. 1995 Sep;45(3):271-81. doi: 10.1016/0306-9877(95)90117-5. PMID 8569551
- [Result] Ter Riet G, de Craen AJM, de Boer A, Kessels AGH. Is placebo analgesia mediated by endogenous opioids? A systematic review. Pain. 1998 Jun;76(3):273-275. doi: 10.1016/S0304-3959(98)00057-8. PMID 9718245
- [Result] Han JS, Terenius L. Neurochemical basis of acupuncture analgesia. Annu Rev Pharmacol Toxicol. 1982;22:193-220. doi: 10.1146/annurev.pa.22.040182.001205. No abstract available. PMID 7044284
- [Derived] Erdogan P, Yardimci H. Analgesic effects of LI4 acupuncture during intrauterine device insertion: a randomized controlled clinical trial. Arch Gynecol Obstet. 2023 Oct;308(4):1361-1368. doi: 10.1007/s00404-023-07106-5. Epub 2023 Jul 19. PMID 37466690